CLINICAL TRIAL: NCT04894032
Title: Postoperative Results of a Meshless Method in the Surgical Treatment of Pelvic Organ Prolapse; Combination of Laparoscopic Uterosacral Ligament and Round Ligament Plication.
Brief Title: Combination of Laparoskopic Uterosacral Ligament and Round Ligament Plication, A Meshless Method in the Surgical Treatment of Pelvic Organ Prolapse.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Zeynep Kamil Maternity and Pediatric Research and Training Hospital (Other)
Responsible Party: Principal Investigator, Sultan Seren Karakus, Specialist, Zeynep Kamil Maternity and Pediatric Research and Training Hospital
Other Study IDs: 9/2021
Record Dates: First submitted 2021-04-05; First posted 2021-05-20 (Actual); Last update posted 2021-05-20 (Actual); Status verified 2021-05

CONDITIONS: Pelvic Organ Prolapse; Prolapse Uterus; Prolapse Bladder
MeSH Terms: conditions — Pelvic Organ Prolapse; Uterine Prolapse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Combination of Laparoscopic Uterosacral Ligament and Round Ligament Plication. — Laparoscopic Uterosacral Ligament Plication, Fixation of PVC fascia and the combination with round ligament plication

SUMMARY:
Postoperative Results of a Meshless Method in the Surgical Treatment of Pelvic Organ Prolapse; Combination of Laparoscopic Uterosacral Ligament and Round Ligament Plication.

DETAILED DESCRIPTION:
Following the approval of the ethics committee, Female patients admitted to Urogynecology and Gynecology Outpatient Clinic of Zeynep Kamil Gynecology and Child Diseases Education and Research Hospital with the complaint of prolapse of the genital organs, who do not respond or not willing to take conservative treatment and have Stage 2 or higher pelvic organ prolapse according to POP-Q staging system and who have completed the fertility period will be included in our study. Patients Age, gravida and parity of the patients, menopausal status, whether she is hysterectomized, the stage of prolapse according to POP-Q and other gynecological examination findings will be recorded.Patients will be asked about preoperative urinary system pathologies (voiding dysfunction, urinary incontinence, recurrent UTI) and Urodynamic examination will be done accordingly.

Prolapsus and its Impact on the quality of life will be recorded preoperatively with quality of life questionnaires.At the early postoperative period and preoperatively, the duration of the operation, blood loss during the surgery, VAS score , and the presence of complications will be recorded. Patients will be called postoperatively for control examination at the 1st month , 6th month , 1st year and subsequently annual control will be done.Objective success; Stage 1 according to POP-Q or no prolapse. Subjective success will be accepted once the patient has no prolapse-related complaints.In the postoperative period, whether there is any change in urinary system and sexual functions will be questioned with the help of questionnaires.Laparoscopic Uterosacral Ligament plication, fixation of PVC fascia and the combination with round ligament plication will be evaluated in terms of efficacy and reliability.

ELIGIBILITY:
Inclusion Criteria:

* Female patients age between 30 to 85
* Having Stage 2 or higher pelvic organ prolapse according to POP-Q staging system
* Patients who accept the surgical treatment

Exclusion Criteria:

* Patients who have a gynecological malignancy
* Pregnant patients

Ages: 30 Years to 85 Years | Sex: Female
Age Groups: Adult, Older Adult
Gender Based: Yes — female patients age between 30 to 85
Study Population: Fmale patients with the complaint of prolapse of the genital organs, who do not respond or not willing to take conservative treatment and have Stage 2 or higher pelvic organ prolapse according to POP-Q staging system and who have completed the fertility period
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2021-01-06 (Actual); Primary Completion 2022-01-06 (Estimated); Study Completion 2022-01-06 (Estimated)

PRIMARY OUTCOMES:
recurrent rate after a meshless method in pelvic prolapse surgery | Through study completion, an average of 6 months
  Combination of Laparoskopic Uterosacral Ligament and Round Ligament plication

CONTACTS AND LOCATIONS:
Locations (1):
- Zeynep Kamil Maternity and Childrens Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No